CLINICAL TRIAL: NCT01109706
Title: Relevance of Plasma PCSK9 Concentration as a Biomarker in Acute Coronary Syndrome.
Acronym: PC-SCA-9
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/10/03-ZE
Record Dates: First submitted 2010-04-20; First posted 2010-04-23 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; PCSK9; cardiovascular safety
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient treated by statines
  Interventions: Other: biological parameters dosage
- patient without normolipidemic treatment
  Interventions: Other: biological parameters dosage

INTERVENTIONS:
Other: biological parameters dosage — 200 patients will be enrolled in the study (n=100 patients under statin treatment, n=100 patients without statin).
  After checking inclusion and non-inclusion criteria and obtaining informed consent from the patients. The SYNTAX score will be calculated and will allow to determine coronary analysis will be done at J1 and J4 (glucose, HbA1C, lipids, ApoA1, ApoB, sterols, plasmatic bile acids, insulinemia, creatinin clearance, hepatic function panel, CRPus and PCSK9 level assessment).
  Then, a sub-group of 30 patients will have supplementary blood analysis at 1 and 6 months after their admission, during their usual follow-up.

SUMMARY:
PCSK9 (Proprotein convertase subtilisin kexin type 9) plays a key role in LDL-cholesterol (LDLC) metabolism by inhibiting LDL receptor (LDLR) at post-transcriptional level. PCSK9 loss of function mutations are associated to decreased LDLC levels and a cardiovascular protection. In this context, the development of pharmacological inhibitors of PCSK9, in association with statins treatment, represents a major therapeutic issue for LDLC modulation. It was previously shown that PCSK9 plasmatic concentration correlated with plasmatic LDLC, TG and glucose concentrations. However, no data are available on predictive value of PCSK9 plasmatic level concerning coronary disease severity.

The main objective of this study is to determine whether plasmatic PCSK9 concentration is linked to coronary damage severity in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion criteria:

* more than 18 years old
* Acute coronary syndrome (ST+ or ST-)
* 2 groups of patients: with statin, and without statin treatment

Exclusion criteria:

* Patient who had cancer during the last 5 years or with cancer in progress
* Patient with severe infection in progress
* Hepatic failure (TP<50%)
* Severe kidney failure
* Patient unable to give his consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes, 18 years old minimum, with an acute coronary syndrome, treated or not with statins, admitted to cardiological intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2011-02-13 (Actual); Primary Completion 2013-09-24 (Actual); Study Completion 2015-07-16 (Actual)

PRIMARY OUTCOMES:
Syntax score (for evaluate coronary damages) and plasmatic concentration of PCSK9 | Day 1, Day 2, Day 3, Day 4
  Assessing the correlation between plasma concentration of PCSK9 and coronary damage severity in patients with acute coronary syndrome. Coronary lesions will be measured using the SYNTAX score (J0: admission day), and PCSK9 concentration will be evaluated using blood analysis (J0 (admission), J1, J2, J3 & J4).

SECONDARY OUTCOMES:
Correlation between PCSK9 and morbidity/mortality | Day 1, Day 2, Day 3, Day 4
  Assessing the correlation between plasma PCSK9 (J1, J2, J3, J4) concentration and one-year morbidity/mortality of patients with acute coronary syndrome
association between PCSK9 and metabolic/inflammatory factors | Day 1, Day 2, Day 3, Day 4
  Identification of metabolic and inflammatory factors (glycemia, insulinemia, HbA1C, CRPus…) associated to plasma PCSK9 concentration
kinetic of PCSK9 for statin-treated patients | Day 1, Day 2, Day 3, Day 4
  Measurement of PCSK9 kinetic variation during ACS acute phase in patients treated with artovastatin 80 mg/day (J1, J2, J3, and J4)
kinetic of PCSK9 after intensive care | Day 1, Day 2, Day 3, Day 4
  Determination of PCSK9 kinetic variation at 1 and 6 months after intensive care, during their normal follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Cariou, MD, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Nantes University hospital, Nantes
  - Nantes University Hospital, Nantes